CLINICAL TRIAL: NCT05143489
Title: The Effect of Pretreatment With Intravenous Lidocaine for Intravenous Contrast: A Double-blinded, Randomized-control Trial
Brief Title: The Effect of Pretreatment With Intravenous Lidocaine for Intravenous Contrast:
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: 1. CTs occur late at night and weekends when their is no availability of the research staff.
  . No activity since a year+
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-01-14
Record Dates: First submitted 2021-11-05; First posted 2021-12-03 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Pain
Keywords: Pain; Pediatrics; Emergency Medicine; Lidocaine
MeSH Terms: conditions — Pain | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preservative Free Lidocaine Group (Active Comparator): The patient will receive a 1mg/kg IV dose of preservative free lidocaine with a max dose of 40mg
  Interventions: Drug: Preservative Free Lidocaine
- Placebo Group (Active Comparator): The patient will receive IV normal saline of 1mg/kg with a max of 40mg
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Preservative Free Lidocaine — The patient will receive a 1mg/kg IV dose of lidocaine with a max dose of 40mg.
  Arms: Preservative Free Lidocaine Group
Drug: Saline — The patient will receive IV normal saline of 1mg/kg with a max of 40mg
  Arms: Placebo Group

SUMMARY:
Intravenous contrast media is commonly used for CT scans for improved image clarity in pediatric emergency medicine. Children who feel discomfort during the administration of IV contrast media may not remain still during the CT scan, which affects the overall study quality and reliability. Therefore, many young patients often undergo procedural sedation in anticipation of movement artifact degrading the diagnostic accuracy. Procedural sedation, while a common procedure in the pediatric emergency department, does have significant complications, and it increases the risk of adverse events for the patient. The risk of airway compromise associated with procedural sedation is particularly concerning in children requiring IV contrast for imaging of an upper airway pathology such as retropharyngeal abscess, as the disease itself narrows the airway. This presents the physician with a dilemma of assessing the extent of the disease without the additional risk of airway compromise by using procedural sedation.Previous research has looked at premedication with steroids prior to IV-contrast media administration to avert an allergic response. However, there has been no investigation of premedication to abate the immediate adverse effects of discomfort associated with IV contrast injection. The safety of IV lidocaine in pediatric patients has been documented in studies of its use for post-operative pain, using doses from 1.0 to 1.5 mg/kg with no known adverse side effects. CT scans with IV contrast are performed on a near-daily basis in the Maimonides pediatric emergency department, usually for the assessment of acute appendicitis. The standard of care in children and adults receiving IV contrast does not include pre-medication to prevent IV contrast-associated discomfort. This double-blinded prospective study aims to determine whether pre-treatment with lidocaine can mitigate the immediate discomfort of IV contrast in verbal children and adolescents who can comply with a pre and post IV contrast pain assessment.

DETAILED DESCRIPTION:
STUDY DESIGN Subjects: Patients aged from 7 to 17 years-old who present to the Maimonides Medical Center's Emergency Department that require a CT scan with IV contrast. Research team members will be notified when the patient requires CT scan with IV contrast and meets the eligibility criteria. Potential subjects will be recruited in the Emergency Department

Eligibility Criteria: Inclusion criteria: Patients with age of 7 to 17 years-old who require a CT scan with IV contrast. Exclusion criteria: Patients with history of seizures, cardiovascular disease, presenting as a trauma, a history of anaphylaxis to lidocaine, or children/adolescents with underlying neurodevelopmental conditions which would interfere with their ability to respond to pre and post IV contrast pain assessments.

Design: This is a prospective, double-blinded randomized control study that will be comparing intravenous lidocaine to a placebo. Patients will be randomized with block randomization. The randomization list will be generated EM Research Manager and given to the EM pharmacist a priori of commencement of the study. The EM Research Manager and EM Pharmacist are not blinded to the study. Once a potential subject has been identified, a member of the research team will obtain consent from the parent or guardian of the subject. The research team member involved with consent and data collection, provider, and subject will all be blinded to which treatment arm they are assigned.

The research team members will monitor each patient and in conjunction with the pharmacy will deliver the assigned treatment to the subject's nurse to administer 10 min prior to the CT scan. If selected for the treatment group, the patient will receive a 1mg/kg IV dose of lidocaine with a max dose of 40mg.15 A patient selected to the control group will an equal volume of normal saline infused. A research team member will be present during the administration of assigned treatment until the completion of the CT scan. The patient will be placed on a cardiopulmonary monitor for the duration of this period. Advanced airway equipment, IV midazolam, and IV intralipids will also be available at bedside during infusion and until completion of CT scan to treat any potential adverse effect associated with lidocaine.

Nominal variables to be collected include gender, chief complaint, pain score at triage, use of pain medication at triage and during the ED course, diagnosis, type of CT scan performed, pre and post-intervention pain score, post-intervention pruritus score, post-intervention burning pain score. The only continuous variable being collected includes age (in years-old).

There will be no interruption or deviation from the standard of clinical care provided to each subject. This study will be run completely in the Pediatric Emergency Department.

Data Collection Procedures: Once a subject has been enrolled, the research team member will review the chart and collect all pertinent information as shown in the data collection template. A questionnaire will be completed prior to administration of the medication as well as following the CT scan which will be administered by the research team member. The investigators will use a combination of the Baker-Wong FACES pain scale and 1 to 10 numerical scale for pain as well as a 5-point Likert scale for discomfort. Once all data has been collected, it will be recorded in password protected document located on a secure server only accessible to members of the research team. All information about the patients will be de-identified. Study investigators will record pain scores, vital signs, and adverse effects at prior to intervention, immediately following intervention, and 15 min following the intervention

The preparing ED pharmacist, research manager, and statistician will be the only ones with knowledge of the study arm to which each participant would be randomized. Treating providers, participants, and the data collecting research team will be blind to the medication route received.

All data will be recorded on data collection sheets, including patients' gender, demographics, medical history, and vital signs, and entered into SPSS (version 27.0; IBM Corp) by the research manager. Development of the randomization list, confirmation of written consent acquisition for all participants, and statistical analyses will be conducted by the research manager and statistician who will work independently of any data collection.

Patients will be closely monitored for any change in vital sings and for adverse effects during the entire study period (up to 120 minutes) by study investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age of 7 to 17 years-old who require a CT scan with IV contrast
* Require CT scan with IV contrast

Exclusion Criteria:

* History of seizures
* Cardiovascular disease
* Presenting as a trauma
* a history of anaphylaxis to lidocaine
* children/adolescents with underlying neurodevelopmental conditions which would interfere with their ability to respond to pre and post IV contrast pain assessments.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rizkalla, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Preservative Free Lidocaine Group | Placebo Group
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preservative Free Lidocaine Group | Placebo Group | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at 15 Minutes Post Medication Administration
Description: We will use a combination of the Baker-Wong FACES pain scale and 1 to 10 numerical scale for pain as well as a 5-point Likert scale for discomfort. Both scales range from no pain to very severe pain with 5 being moderate pain.
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preservative Free Lidocaine Group | Placebo Group
Number analyzed (Participants) | 1 | 2
score on a scale | 0 (0) | 0 (0)

2. Primary Outcome: Pain Score at 30 Minutes Post Medication Administration
Description: as for outcome 1
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preservative Free Lidocaine Group | Placebo Group
Number analyzed (Participants) | 1 | 2
score on a scale | 0 (0) | 3.50 (4.95)

3. Secondary Outcome: Pain Score at 60 Minutes Post Medication Administration
Description: as for outcome 1
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preservative Free Lidocaine Group | Placebo Group
Number analyzed (Participants) | 1 | 2
score on a scale | 0 (0) | 3.0 (4.24)

4. Secondary Outcome: Pain Score at 90 Minutes Post Medication Administration
Description: as for outcome 1
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preservative Free Lidocaine Group | Placebo Group
Number analyzed (Participants) | 1 | 2
score on a scale | 0 (0) | 2 (2.83)

5. Secondary Outcome: Pain Score at 120 Minutes Post Medication Administration
Description: as for outcome 1
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Preservative Free Lidocaine Group | Placebo Group
Number analyzed (Participants) | 1 | 2
score on a scale | 0 (0) | 4 (5.66)

ADVERSE EVENTS:
Time Frame: 120 minutes
Arm/Group | Preservative Free Lidocaine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT05143489/Prot_SAP_000.pdf